CLINICAL TRIAL: NCT02313415
Title: Clinical Study of the Treatment of Infertility Caused by Recurrent Intrauterine Adhesions by Collagen Scaffold Loaded With Umbilical Cord -Derived Mesenchymal Stem Cells (UC-MSCs)
Brief Title: Treatment of Infertility by Collagen Scaffold Loaded With Umbilical Cord Derived Mesenchyma Stem Cells
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Collaborators: Institute of genetic development, Chinese Academy of Sciences (Unknown); Institute of Zoology, Chinese Academy of Sciences (Other Government)
Responsible Party: Principal Investigator, Yali Hu, MD,PhD, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20141206
Record Dates: First submitted 2014-12-07; First posted 2014-12-10 (Estimated); Last update posted 2017-10-24 (Actual); Status verified 2017-10

CONDITIONS: Infertility; Intrauterine Adhesions
MeSH Terms: conditions — Infertility; Gynatresia

STUDY DESIGN:
Intervention Model Description: treatment of infertility caused by recurrent intrauterine adhesions by collagen scaffold loaded with UC-MSCs
Oversight: Data Monitoring Committee: No

ARMS (1):
- UC-MSCs therapy (Experimental): transplant collagen scaffold loaded with UC-MSCs to treat infertility caused by recurrent intrauterine adhesions
  Interventions: Procedure: UC-MSCs therapy

INTERVENTIONS:
Procedure: UC-MSCs therapy — Before considering whether patients meet the inclusion criteria, they are diagnosed as intrauterine adhesions with at least one unsuccessful hysteroscopic surgery. And after that there will be history taking, physical examination, ultrasound examination and hysteroscopy examination. If they agree to participate, they will receive separation of adhesions by hysteroscopy surgery and endometrial biopsies, then a collagen scaffold loaded with UC-MSCs will be transplanted into the uterine cavity. The procedure was performed after taking 6 mg/day × 10 days Progynova, continuous administration of the same dosage Progynova for 30 days and 60mg of progesterone were injected on the 30th day post-operation. Postoperative observation including ultrasound examination once a month for 3 times and hysteroscopy after 3 months. The doctor will select an appropriate time for pregnancy and follow-up including requiring patients to do some unscheduled visits.

SUMMARY:
Study of the treatment of infertility caused by recurrent intrauterine adhesions (IUA) by collagen scaffold loaded with umbilical cord derived mesenchymal stem cells (UC-MSCs) to provide clinical evidence of safety and effectiveness for the treatment of uterine infertility.

DETAILED DESCRIPTION:
Infertility is defined as a women fails to become pregnant after having a normal sex life for two years without contraception. There is limited treatment to the infertility caused by severe IUA especially recurrent IUA after adhesiolysis which hinders embryos implantation. The existing drugs, physical or surgical treatments had no significant effects to severe recurrent intrauterine adhesions. Collagen is the main component of the extracellular matrix with good biocompatibility, UC-MSCs have been used in the clinical treatment of diseases, and achieved good results. In this study, collagen scaffold and umbilical cord blood-derived mesenchymal stem cells are combined, and they showed good biological safety.

ELIGIBILITY:
Inclusion Criteria:

* Secondary infertility or failure of embryo transfer caused by recurrent intrauterine adhesions who desired to be pregnant
* Hysteroscopy examination confirmed intrauterine adhesions
* Sign a consent form
* Follow the test plan and follow-up process

Exclusion Criteria:

* have hysteroscopic contraindications
* Chromosome karyotype abnormalities
* Congenital uterine malformations
* Severe adenomyosis
* Contraindications to estradiol treatment
* Medical history of pelvic tumors or receiving pelvic radiotherapy

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2014-11-28 (Actual); Primary Completion 2015-01-28 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
live birth rate | 30 months
  A baby born alive after 20 weeks gestation was classified as a live birth.

SECONDARY OUTCOMES:
Reduction of intrauterine adhesion | 3 months post-surgery
  Hysteroscopic inspection to verify degree of adhesion
The change of endometrial thickness | up to 3 months
  Measure the endometrial thickness during late proliferating phase by ultrasound
ongoing pregnant rate | 30 months
  The presence of at least one fetus with heart pulsation on ultrasound beyond 8 weeks

OTHER OUTCOMES:
The change of menstrual blood volume | baseline and 1 month
  Understanding the menstrual blood volume after surgery comparing with pre-operation.

CONTACTS AND LOCATIONS:
Overall Officials: Yali HU, MD,PhD, Principal Investigator — Vice-president of the Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Locations (1):
- Nanjing Drum Tower Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cao Y, Sun H, Zhu H, Zhu X, Tang X, Yan G, Wang J, Bai D, Wang J, Wang L, Zhou Q, Wang H, Dai C, Ding L, Xu B, Zhou Y, Hao J, Dai J, Hu Y. Allogeneic cell therapy using umbilical cord MSCs on collagen scaffolds for patients with recurrent uterine adhesion: a phase I clinical trial. Stem Cell Res Ther. 2018 Jul 11;9(1):192. doi: 10.1186/s13287-018-0904-3. PMID 29996892